CLINICAL TRIAL: NCT01704963
Title: A Phase 1 Study of the Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 in Subjects With Recurrent Mature B-Cell Neoplasms
Brief Title: A Study to Evaluate the Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 in Patients With Recurrent Mature B-Cell Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100896; PCI-32765-JPN-101 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Recurrent Mature B-cell Neoplasms
Keywords: Recurrent mature B-cell neoplasms; B-cell malignancies; Bruton's Tyrosine Kinase (Btk) Inhibitor; PCI-32765; Tumor; Pharmacokinetics; Japanese
MeSH Terms: conditions — Neoplasms | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- PCI-32765 (Experimental): Patients will receive oral doses of PCI-32765 in Cohort 1, Cohort 2 and CLL/SLL Cohort. In Cohort 1, single oral dose of PCI-32765 140 mg and 280 mg will be given before administration of daily oral doses of 420 mg per day for 35 days in Cycle 1 and for 28 days in Cycle 2 and thereafter. In Cohort 2 and CLL/SLL Cohort, PCI-32765 560 mg and 420 mg per day, respectively will be administered daily for 35 days in Cycle 1 and for 28 days in Cycle 2 and thereafter.
  Interventions: Drug: PCI-32765

INTERVENTIONS:
Drug: PCI-32765 — PCI-32765 will be administered in Cohort 1, Cohort 2 and CLL/SLL Cohort. In Cohort 1, single oral dose of PCI-32765 140 mg and 280 mg will be administered before daily oral doses of 420 mg per day for 35 days in Cycle 1 and for 28 days in Cycle 2 and thereafter. In Cohort 2 and CLL/SLL Cohort, PCI-32765 560 mg and 420 mg per day, respectively will be administered daily for 35 days in Cycle 1 and for 28 days in Cycle 2 and thereafter.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 in Japanese patients with recurrent mature B-cell neoplasms.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (study conducted at multiple sites), dose escalation study. The study consists of 3 phases, including, the screening phase (within 14 days prior to the first study medication), the treatment phase, and the follow up phase. In the treatment phase, patients with recurrent mature B-cell neoplasms will be divided into 2 cohorts: Cohort 1 (consisting of between 3 and 12 patients), and Cohort 2 (consisting of between 6 and 12 patients). Cohort 1 will be further divided into 2 phases: a single dose (SD) phase and a multiple dose (MD) phase. During the initial SD phase, patients will first receive a single dose of PCI-32765 at 140 mg. After a washout period (period when the participant is not receiving any study medication) of between 72 and 168 hours, patients will then receive a second single dose of PCI-32765 at 280 mg. Following a second washout period, patients will enter the MD phase, where they will receive PCI-32765 at multiple doses of 420 mg per day for 35 days during the first cycle (35 days in Cycle 1) and for 28 days during the second cycle (28 days in Cycle 2) and every cycle thereafter. In cohort 2, patients will receive multiple doses of 560 mg per day for 35 days in Cycle 1, 28 days in Cycle 2, and every cycle thereafter. The patient's registration in Cohort 2 will be started after tolerability of Cohort 1 is confirmed. Tolerability of each dose level will be evaluated based on the dose-limiting toxicity (DLT) occurrence rate in Cycle 1 of each Cohort. Following the tolerability of the 420 mg/day dose level in subjects with mature B-cell neoplasms is confirmed in Cohort 1, a CLL/SLL Cohort will be added to further evaluate the safety and tolerability of this dose in this specific population in Japanese since 420 mg/day is the globally recommended dose for subjects with CLL and SLL, which are specific disease entities within mature B-cell neoplasms. Between 6 and 12 subjects will be enrolled in the CLL/SLL Cohort and will receive continuous dosing of PCI-32765 at 420 mg/day for 35 days in Cycle 1 and for 28 days in Cycle 2 and thereafter. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, and corneal eye examination will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have body weight at least 40 kilogram (kg)
* Patients with recurrent mature B-cell neoplasms as defined according to WHO classification, including small lymphocytic lymphoma/ chronic lymphocytic leukemia, mantle cell lymphoma, and follicular lymphoma
* Have measurable disease [for Non-Hodgkin's Lymphoma (NHL) bi-dimensional disease more than or equal to 2 cm diameter in at least one dimension and for chronic lymphocytic leukemia more than or equal to 5000 leukemia cells/cubic mm]
* Have failed more than or equal to 1 previous treatment and no standard therapy is available
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Patients with plasma cell neoplasm as defined according to WHO classification
* Patients who have received prior allogeneic hematopoietic stem cell transplant
* Patients who have received immunotherapy, chemotherapy, radiotherapy or experimental therapy within 4 weeks before first day of study medication
* Past history of major surgery within 4 weeks before the first day of study medication
* Patients with central nervous system involvement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Screening (Day -14) to until 30 days after the last dose

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to the time of the last measurable concentration (AUClast) | Days 1-2, 8-9, 15, 22 and 29 during Cycle 1 of each cohort
  Pharmacokinetic parameter AUClast of PCI-32765 and its metabolite PCI-45227 will be measured when PCI-32765 is administered daily as oral doses in each cohort.
Area under the plasma concentration-time curve from time 0 to infinity time (AUC∞) | Days 1-2, 8-9, 15, 22 and 29 during Cycle 1 of each cohort
  Pharmacokinetic parameter AUC∞ of PCI-32765 and its metabolite PCI-45227 will be measured when PCI-32765 is administered daily as oral doses in each cohort.
Maximum plasma concentration (Cmax) | Days 1-2, 8-9, 15, 22 and 29 during Cycle 1 of each cohort
  Pharmacokinetic parameter Cmax of PCI-32765 and its metabolite PCI-45227 will be measured when PCI-32765 is administered daily as oral doses in each cohort.
Time to reach maximum plasma concentration (tmax) | Days 1-2, 8-9, 15, 22 and 29 during Cycle 1 of each cohort
  Pharmacokinetic parameter tmax of PCI-32765 and its metabolite PCI-45227 will be measured when PCI-32765 is administered daily as oral doses in each cohort.
Terminal elimination half-life (t1/2) | Days 1-2, 8-9, 15, 22 and 29 during Cycle 1 of each cohort
  Pharmacokinetic parameter t1/2 of PCI-32765 and its metabolite PCI-45227 will be measured when PCI-32765 is administered daily as oral doses in each cohort.
Pharmacodynamic evaluations | Days 1-2, 8-9, 15, and 29 during Cycle 1, and on Days 1 and 15 during Cycle 3, 5, 7, 9, and 11 of each cohort
  Pharmacodynamic evaluations of PCI-32765 will be conducted under supervision by collecting venous blood samples.
Tumor response | Days 22 to 28 of Cycles 2, 4, 6, and every even-numbered cycle thereafter
  Patients will be evaluated for tumor response according to the International Working Group (IWG) Revised Criteria for Malignant Lymphoma or the Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (4):
- Japan (4):
  - Kyoto
  - Nagoya
  - Sendai
  - Tokyo

REFERENCES:
- [Result] Tobinai K, Ogura M, Ishizawa K, Suzuki T, Munakata W, Uchida T, Aoki T, Morishita T, Ushijima Y, Takahara S. Safety and tolerability of ibrutinib monotherapy in Japanese patients with relapsed/refractory B cell malignancies. Int J Hematol. 2016 Jan;103(1):86-94. doi: 10.1007/s12185-015-1900-3. Epub 2015 Nov 20. PMID 26588924
- See also: A Phase 1 Study of the Bruton's Tyrosine Kinase (Btk) Inhibitor PCI-32765 in Subjects With Recurrent Mature B-Cell Neoplasms — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3564&filename=CR100896_CSR.pdf